CLINICAL TRIAL: NCT05266066
Title: Multicenter Randomized Clinical Trial of Antimicrobial Treatment in Ventilator-associated Tracheobronchitis
Brief Title: Ventilator-associated Tracheobronchitis Initiative to Conduct Antibiotic Evaluation
Acronym: VATICAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Hospital Israelita Albert Einstein (Other); Hospital do Coracao (Other); Hospital Moinhos de Vento (Other); Hospital Alemão Oswaldo Cruz (Other); BP - A Beneficência Portuguesa de São Paulo (Unknown); Brazilian Research in Intensive Care Network (BRICNet) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48749421.0.1001.5461
Record Dates: First submitted 2022-02-15; First posted 2022-03-04 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Ventilator Associated Tracheobronchitis; Tracheobronchitis
Keywords: Antibiotics; Ventilator associated Tracheobronchitis; Mechanical ventilation; Critically ill
MeSH Terms: conditions — Critical Illness | interventions — Watchful Waiting; Anti-Infective Agents

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to Clinical observation without antibiotic therapy for VAT vs. 7 day antibiotic course.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical observation without antibiotic therapy for VAT (Experimental): Patients will receive standard care and no antibiotic therapy for VAT. Antibiotics will be prescribed if other infections and/or organ dysfunction ensues (especially shock) or there is progression to pneumonia
  Interventions: Other: Clinical observation without antibiotic therapy for VAT
- 7 day antibiotic course for VAT (Active Comparator): Patients will receive standard care and 7 day course of antibiotic therapy for VAT.
  Interventions: Other: 7 day antibiotic course for VAT

INTERVENTIONS:
Other: Clinical observation without antibiotic therapy for VAT — Patients will receive standard care plus antibiotic if new organ dysfunction or new infections other than VAT.
  Arms: Clinical observation without antibiotic therapy for VAT
Other: 7 day antibiotic course for VAT — Patients will receive standard care plus 7 day course of antibiotic.
  Arms: 7 day antibiotic course for VAT

SUMMARY:
The Ventilator Associated tracheobronchitis Initiative to Conduct Antibiotic evaluation (VATICAN) trial is a national, multicenter, non-inferiority trial in ICU patients comparing antibiotic treatment for 7 days versus clinical observation without antibiotic treatment for patients with ventilator-associated tracheobronchitis.

DETAILED DESCRIPTION:
There is no consensus on the need for antibiotic treatment for ventilator-associated tracheobronchitis (VAT). There's a lack of high-quality clinical data on this subject, and although some observational studies recommend antibiotic treatment for VAT, some guidelines do not. The VATICAN is a prospective, randomized, single-blinded (analysis), non-inferiority trial evaluating antibiotic treatment for patients with ventilator-associated tracheobronchitis. Patients with clinically diagnosed tracheobronchitis will be randomized to receive antibiotics for 7 days versus clinical observation without antibiotic treatment for VAT. The primary hypothesis is that clinical observation without antibiotic treatment is noninferior to 7-day antibiotic course.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the participating ICUs
* Invasive Mechanical ventilation ≥ 48 hours
* Available chest imaging of screening day
* Clinical diagnosis of VAT, defined by the presence of:

  1. Temperature >38.0°C or <36°C OR leukocytes >12000/mL or <4000/mL or presence >10% of immature forms, AND
  2. Onset of purulent tracheal secretion, or change in characteristics of the secretion, or increase in the amount of respiratory secretion, or increased need for aspiration
* Culture of tracheal secretion from the day of screening under analysis or collected for analysis

Exclusion Criteria:

* Pregnant or lactating women
* Indication of use of antibiotics or use of systemic antibiotics for any indications at the time of screening
* Hemodynamic instability, defined as hypotension unresponsive to volume expansion or increase in vasopressor dose > 0.1mcg/kg/min of noradrenaline or equivalent in the past 6 hours
* Worsening of gas exchange, defined as an increase in the fraction of inspired oxygen ≥ 20% or an increase in positive end-expiratory pressure (PEEP) ≥ 3 cm of water after a stability period ≥ 2 days
* Prolonged mechanical ventilation, defined by use of invasive mechanical ventilation for 21 days or more
* Presence of pulmonary radiological image suggestive of new infectious infiltrate
* Previous lung disease that makes radiological interpretation for the diagnosis of VAP difficult
* Previous diagnosis of ventilator associates pneumonia (VAP) during hospitalization
* Neutropenic patients (neutrophils <1000/mL)
* Known severe immunosuppression
* Tracheostomized patients at the time of screening
* Inclusion in the study in the past 30 days
* Expected limitation of care or early withdrawal of supportive therapies (< 7 days)
* Patients with a survival expectancy of less than 48 hours
* Refusal of consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Ventilator free days | 28 days after randomization
  Days alive and free from mechanical ventilation

SECONDARY OUTCOMES:
Ventilator associated pneumonia-free survival (Key secondary outcome) | 28 days after randomization
  The time between randomization and the diagnostic event of ventilator associated pneumonia or death
Mortality | 28 days after randomization
  All cause mortality
Ventilator associated pneumonia | 14 and 28 days after randomization
  Ventilator associated pneumonia incidence
Intensive care unit free days | 28 days after randomization
  Days alive and free from intensive care unit
Organ dysfunction | Between randomization and day 7.
  Variation in organ dysfunction (measured by the Sequential Organ Failure Assessment Score). Sequential Organ Failure Assessment scores are measured in 6 organ systems (cardiovascular, hematologic, gastrointestinal, renal, pulmonary and neurologic), with each organ scored from 0 to 4, resulting in an aggregated score that ranges from 0 to 24, with higher scores indicating greater dysfunction.
Microbiological isolation of multi-resistant bacteria | 28 days after randomization
  Microbiological isolation of multi-resistant bacteria. Any isolation of by microbiological cultures of multi-resistant bacteria following the definition:
  Acinetobacter baumannii: Resistant to carbapenems and/or polymyxins Pseudomonas aeruginosa: Resistant to carbapenems and/or polymyxins Enterobacteriaceae: Resistant to carbapenems and/or polymyxins (in enterobacteria naturally sensitive to polymyxins) Vancomycin-resistant Enterococcus faecium (VRE) Methicillin/Oxacillin Resistant Staphylococcus aureus (MRSA) Methicillin/Oxacillin-Resistant Coagulase Negative Staphylococcus (MRSA)
Antibiotic free days | 28 days after randomization
  Days alive and free from antibiotic
Cost analysis | For the first 28 days after randomization
  Cost effectiveness analysis. Direct and indirect hospital costs will be measured and used in the analyses. For that, a local costing system will be built, using the absorption costing methodology (top-down).

OTHER OUTCOMES:
Nosocomial infections | 28 days after randomization
  Incidence of culture positive nosocomial infections in 28 days
Adverse events | 28 days after randomization
  Severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bruno M Tomazini, MD, Principal Investigator — Hospital Sírio-Libanês
Locations (16):
- Brazil (16):
  - Hospital OTOClinica, Fortaleza, Ceará
  - Hospital Vila Velha, Vila Velha, Espírito Santo
  - Hospital Santa Casa de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Vila da Serra, Nova Lima, Minas Gerais
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital São Joao Del Rei, São João del Rei, Minas Gerais
  - Hospital Universitário Regional do Norte do Paraná, Londrina, Paraná
  - Hospital Municipal de Maringá, Maringá, Paraná
  - Hospital Tricentenário, Olinda, Pernambuco
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Hospital Itapetininga, Itapetininga, São Paulo
  - Hospital Unimed Limeira, Limeira, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - Hospital Samaritano, São Paulo, São Paulo
  - Hospital São Paulo, São Paulo, São Paulo
  - Hospital Santa Casa de Sorocaba, Sorocaba, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) might be shared upon request and approval by the study committee after the study completion.
Supporting Information: Study Protocol, SAP
Time Frame: One year after study completion.
Access Criteria: Individual patient data might be shared upon request and approval by the study committee after the study completion.

REFERENCES:
- [Background] IMPACTO-MR, VATICAN Trial Investigators and BRICNet; Tomazini BM, Besen BAMP, Dietrich C, Gandara APR, Silva DP, Pinheiro CCG, Luz MN, Mattos RR, Reis LFL, Roepke RML, Duarte CSLG, Nassar Junior AP, Veiga VC, Arns B, Nascimento GM, Pereira AJ, Cavalcanti AB, Machado FR, Azevedo LCP. VATICAN (Ventilator-Associated Tracheobronchitis Initiative to Conduct Antibiotic Evaluation): protocol for a multicenter randomized open-label trial of watchful waiting versus antimicrobial therapy for ventilator-associated tracheobronchitis. Crit Care Sci. 2024 Aug 26;36:e20240029en. doi: 10.62675/2965-2774.20240029-en. eCollection 2024. PMID 39194024
- [Background] Tomazini BM, Nassar AP Jr, Lisboa TC, Azevedo LCP, Veiga VC, Catarino DGM, Fogazzi DV, Arns B, Piastrelli FT, Dietrich C, Negrelli KL, Jesuino IA, Reis LFL, Mattos RR, Pinheiro CCG, Luz MN, Spadoni CCDS, Moro EE, Bueno FR, Sampaio CSJC, Silva DP, Baldassare FP, Silva ACA, Veiga T, Barbante L, Lambauer M, Campos VB, Santos E, Santos RHN, Laranjeiras LN, Valeis N, Santucci E, Miranda TA, Patrocinio ACLD, Carvalho A, Sousa EMC, Sousa AHF, Malheiro DT, Bezerra IL, Rodrigues MB, Malicia JC, Silva SSD, Gimenes BDP, Sesin GP, Zavascki AP, Sganzerla D, Medeiros GS, Santos RDRMD, Silva FKR, Cheno MY, Abrahao CF, Oliveira Junior HA, Rocha LL, Nunes Neto PA, Pereira VC, Paciencia LEM, Bueno ES, Caser EB, Ribeiro LZ, Fernandes CCF, Garcia JM, Silva VFF, Santos AJD, Machado FR, Souza MA, Ferronato BR, Urbano HCA, Moreira DCA, Souza-Dantas VC, Duarte DM, Coelho J, Figueiredo RC, Foreque F, Romano TG, Cubos D, Spirale VM, Nogueira RS, Maia IS, Zandonai CL, Lovato WJ, Cerantola RB, Toledo TGP, Tomba PO, Almeida JR, Sanches LC, Pierini L, Cunha M, Sousa MT, Azevedo B, Dal-Pizzol F, Damasio DC, Bainy MP, Beduhn DAV, Jatoba JDVN, Moura MTF, Rego LRM, Silva AVD, Oliveira LP, Sodre Filho ES, Santos SSD, Neves IL, Leao VCA, Paes JLL, Silva MCM, Oliveira CD, Santiago RCB, Paranhos JLDR, Wiermann IGDS, Pedroso DFF, Sawada PY, Prestes RM, Nascimento GC, Grion CMC, Carrilho CMDM, Dantas RLAM, Silva EP, Silva ACD, Oliveira SMB, Golin NA, Tregnago R, Lima VP, Silva KGND, Boschi E, Buffon V, Machado AS, Capeletti L, Foernges RB, Carvalho AS, Oliveira Junior LC, Oliveira DC, Silva EM, Ribeiro J, Pereira FC, Salgado FB, Deutschendorf C, Silva CFD, Gobatto ALN, Oliveira CB, Dracoulakis MDA, Alvaia NOS, Souza RM, Araujo LLC, Melo RMV, Passos LCS, Vidal CFL, Rodrigues FLA, Kurtz P, Shinotsuka CR, Tavares MB, Santana IDV, Gavinho LMDS, Nascimento AB, Pereira AJ, Cavalcanti AB. IMPACTO-MR: a Brazilian nationwide platform study to assess infections and multidrug resistance in intensive care units. Rev Bras Ter Intensiva. 2022 Oct-Dec;34(4):418-425. doi: 10.5935/0103-507X.20220209-pt. Epub 2023 Mar 3. PMID 36888821